CLINICAL TRIAL: NCT03742570
Title: The Turkish Version of The Childhood Bladder and Bowel Dysfunction Questionnaire (CBBDQ): Cross-Cultural Adaptation, Reliability and Construct Validity
Brief Title: Turkish Version of Childhood Bladder and Bowel Dysfunction Questionnaire
Status: Completed | Type: Observational
Sponsor: Okan University (Other)
Responsible Party: Principal Investigator, Gamze Tosun Aydin, Principal Investigator, Okan University
Other Study IDs: OkanUn
Record Dates: First submitted 2018-11-04; First posted 2018-11-15 (Actual); Last update posted 2018-11-19 (Actual); Status verified 2018-11

CONDITIONS: Children
Keywords: Childhood Bladder and Bowel Dysfunction Questionnaire; Reliability; Turkish

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CBBDQ: A Questionnaire
  Interventions: Behavioral: CBBDQ

INTERVENTIONS:
Behavioral: CBBDQ — a questionnaire for childood bladder and bowel dysfunctions

SUMMARY:
Objectives:The aim of this study was to translate the Childhood Bladder and Bowel Dysfunction Questionnaire into Turkish, adapt it for use with parents of 5-12 year old children and determine the reliability and construct validity of the Turkish version. The main hypothesis of our study was that it would be possible to translate and culturally adapt the CBBDQ into a Turkish version, so that Turkish parents could understand it. Additionally, we hypothesized that the Turkish version would provide adequate internal consistency and test-rest reliability and acceptable construct validity.

Methods:The Childhood Bladder and Bowel Dysfunction Questionnaire was guideline driven translated into Turkish and administered twice, at 7-day intervals, to parents of children to assess test-retest reliability. Cronbach's α was used for internal consistency and the inter-rater correlation coefficient was used to calculate test-retest reliability. The Dysfunctional Voiding and Incontinence Scoring System (DVISS) and Pediatric Quality of Life Inventory (PedsQL) in 5-7, 8-12 years old children were used as an external criterion to estimate construct validity.

DETAILED DESCRIPTION:
The study was conducted as a questionnaire-based cross-sectional survey of parents of children (5-12y) with urinary incontinence, enuresis, constipation/fecal incontinence in two phases.

Phase 1: Translation Process & Cultural Adaptation. The CBBDQ was translated into Turkish and culturally adapted in accordance with the stages recommended by Beaton.

Phase 2: Field Testing Prior to inclusion, the parents completed an informed consent form, which had been approved by the ethical committee at Istanbul University (IRB study protocol: 2017/487).

Inclusion criteria were: 1) parents of children, aged between 5 to 12 years; 2) whose children suffered from urinary incontinence, enuresis nocturia, constipation/fecal incontinence; and 3) parents and children read and approved the informed consent form. Exclusion criteria were: 1) the presence of urinary tract infection; 2) patients having spinal cord injury or neurological disease; 3) not being able to communicate.

The parents of children were asked to complete the Turkish version of the CBBDQ and the previously validated Turkish version of the DVISS and the Parent-Proxy-Report of the PedsQL (5-7, 8-12) (12, 13). The physiotherapist distributed the Turkish CBBDQ, the DVISS and the PedsQL (5-7, 8-12) to the parents in the waiting room after an interview with the psychiatrist. The parents were then asked to complete the Turkish-CBBDQ5-12y by telephone, 7 days after their first assessment, to determine the test-retest reliability by the same physiotherapist. After parents completed the questionnaire, the physical therapists checked for missing responses. The parents who skipped a question on the questionnaire were asked to give the reason for this. Any difficulty in understanding the question or incompatibility with their problem was noted.

Reported Outcome Measures The CBBDQ consists of two subscales: (1) the bladder symptoms scale (10 items) and (2) the bowel symptoms scale, including abdominal pain and bloated belly (8 items). The parents were asked to indicate the presence of the symptoms applying the past months, using a 5-point Likert scale by checking a box labelled 0-4. '0' means no, '4' means almost every day or every day.

The DVISS is a 14-item questionnaire originally designed in Turkish with the aim to diagnose patients with dysfunctional voiding. The DVISS includes 12 questions on bladder dysfunction, one on bowel dysfunctions and one on quality of life and has variable (Likert scales, dichotomous) answering options. The total score ranged from 0 to 35 points; sum scores higher from 9 points indicate increased disease severity.

The PedsQL measurement model is a modular approach to assess health-related quality of life in healthy children and adolescents and those with acute and chronic health conditions. This scale was developed for children between 5-7 years of age and 8-12 years of age and their parents. In the 5-7-year age group, the questionnaire is filled in by the researcher with the help of a diagram that symbolizes facial expressions of the child like happy, neutral or sad. Unlike other age groups, the response scale of the child's form has three options. There is a parent and child form for the 8-12 age group. Scores of 23 items are scored in 3 areas. First, the total score of the scale is calculated as the sum of all the items over the items answered on all the scales. Second is the physical health total score, and third is the total score of psychosocial health which is calculated by evaluating sum of the item scores emotional, social and school functioning (14). The items are scored between 0-100 points. If the answer to the question is never it is marked as 0 = 100 points, rarely is marked as 1 = 75, sometimes is marked as 2 = 50, frequently is marked as 3 = 25, and almost always is marked as 4 = 0. The points are divided into the total answer number of questions. If more than 50% of the questions are missing, the score cannot be evaluated. The higher the PedsQL total score, the better perceived health-related quality of life.

Statistical Analysis All statistical analyses were performed with the Statistical Package for the Social Sciences (SPSS) 17.5 (SPSS Inc., Chicago, IL, USA). A P-value < 0.05 was considered to indicate statistical significance. We performed a power analysis to determine sample size at the beginning of the study. To achieve an Intraclass Correlation Coefficient (ICC) of at least 0.8 a sample size of 50 participants was needed. For the descriptive analyses, data are expressed as means and standard deviations for continuous variables or as frequencies and percentages for categorical variables and the dispersion/distribution (standard deviations, ranges) for continuous variables. The Kolmogorov - Smirnov test was used to assess the normality of the distribution of scores. Internal consistency, test-retest reliability, construct validity, and ceiling and floor effects were analyzed in this study.

Reliability Reliability refers to the consistency of measurement and includes internal consistency as well as the test-retest reliability. A measure of the homogeneity of the questions within a questionnaire (internal consistency) was calculated by using coefficient of Cronbach's alpha. An α of 0.7 is considered fair, 0.8 is good, and 0.9 represents excellent internal consistency. In this study, baseline data were used to assess the internal consistency of the Turkish version of the-CBBDQ.

The test-retest reliability represents a scale's effectiveness in producing consistent results when administered on different days when an individual's status has remained stable. The outcome measure was applied and then re-applied after 7 days. The results were then compared for agreement by means of an intra-class correlation coefficient (ICC), which was used to measure the test-retest reliability of the Turkish-CBBDQ5-12y. The ICC was also used to calculate standard error measurement (SEM), which is an index of measurement precision. The SEM is calculated as the standard deviation (SD) of the scores the square root of (1-ICC). The minimal detectable change (MDC) refers to the minimal amount of change within the measurement error. The SEM was used to determine the minimum detectable change at the 95% limit of confidence (MDC 95%) and was calculated as the SEM times 1.96 times the square root of 2.

Construct Validity Validity refers to the degree to which a study accurately reflects or assesses the specific concept that the researcher is attempting to measure. In this study, we examined three aspects of validity: construct (convergent and divergent) validity. Evidence for construct validity of the Turkish version of the CBBDQ will be tested by determining its relationship with the Turkish version of DVISS and the PedsQL (5-7, 8-12). The DVISS was used to assess the convergent validity. Evidence for divergent validity was provided by determining the relationships with the PedsQL (5-7, 8-12). Spearman correlation coefficients and their 95% confidence intervals were calculated to assess construct validity. Correlation values are rated as: r ≥ 0.81-1.0 is excellent; 0.61-0.80, very good; 0.41-0.60, good; 0.21-0.40, fair; and 0.00-0.20, poor).

Distribution and Ceiling/Floor Effects Ceiling and floor effects of the Turkish-CBBDQ at the first and second tests were assessed by calculating the proportion of the patients scoring the maximum (72) or minimum (0) scores relative to the total number of patients. Descriptive statistics (number of percentage) were calculated to determine distribution and ceiling/floor effects, which were considered to be relevant if more than 30% of the subjects experienced them.

ELIGIBILITY:
Inclusion Criteria:

* parents of children, aged between 5 to 12 years;
* whose children suffered from urinary incontinence, enuresis nocturia, constipation/fecal incontinence;
* parents and children read and approved the informed consent form.

Exclusion Criteria:

* the presence of urinary tract infection;
* patients having spinal cord injury or neurological disease;
* not being able to communicate.

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The study was conducted as a questionnaire-based cross-sectional survey of parents of children (5-12y) with urinary incontinence, enuresis, constipation/fecal incontinence.
Sampling Method: Probability Sample
Enrollment: 85 (Actual)
Dates: Start 2016-04-13 (Actual); Primary Completion 2018-06-15 (Actual); Study Completion 2018-10-15 (Actual)

PRIMARY OUTCOMES:
DVISS | 2017-2018
  The DVISS is a 14-item questionnaire originally designed in Turkish with the aim to diagnose patients with dysfunctional voiding. The DVISS includes 12 questions on bladder dysfunction, one on bowel dysfunctions and one on quality of life and has variable (Likert scales, dichotomous) answering options. The total score ranged from 0 to 35 points; sum scores higher from 9 points indicate increased disease severity

CONTACTS AND LOCATIONS:
Overall Officials: Gamze Aydin, MSc, Principal Investigator — Okan University

IPD SHARING:
Plan to Share IPD: No